CLINICAL TRIAL: NCT02648945
Title: A Comparative Study Between Effects of Low and High Intensity Exercise in Improving Working Memory Among Students With Anxiety Symptoms
Brief Title: Effects of Low and High Intensity Exercise in Improving Working Memory Among Students With Anxiety Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Manisha Parai (Other)
Collaborators: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Sponsor-Investigator, Manisha Parai, Lecturer, Universiti Tunku Abdul Rahman
Organization: Universiti Tunku Abdul Rahman (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U/SERC/86/2015
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Aerobic Exercise
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- high intensity exercise (Active Comparator): high intensity exercise on a treadmill according to Balke's Protocol.
  high intensity of exercises for each group of 15 participants were set at 80-85% VO2 max (Schneider, S., et al., 2009). To determine the targeted HR for low and high intensity aerobic exercise for each participant, the needed VO2 max percentages were subbed into the Swain equation as follows: %VO2 max = (%HRmax - 37)/0.64 Exercise HR/HRmax = %HRmax
  After rearrangement, it will be:
  %HRmax = %VO2 max x 0.64 + 37 Exercise HR = %HRmax x HRmax During the experimental session, each participant performed physical exercise training on the treadmill according to Balke's Protocol. The reliability of this protocol was tested by Leddy, et. al. (2011).
  Interventions: Other: Exercise
- low intensity exercise (Active Comparator): low intensity exercise on a treadmill according to Balke's Protocol. low intensity of exercises for each group of 15 participants were set at 50-55% VO2 max (Schneider, S., et al., 2009). To determine the targeted HR for low and high intensity aerobic exercise for each participant, the needed VO2 max percentages were subbed into the Swain equation as follows: %VO2 max = (%HRmax - 37)/0.64 Exercise HR/HRmax = %HRmax
  After rearrangement, it will be:
  %HRmax = %VO2 max x 0.64 + 37 Exercise HR = %HRmax x HRmax During the experimental session, each participant performed physical exercise training on the treadmill according to Balke's Protocol. The reliability of this protocol was tested by Leddy, et. al. (2011).
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — first, Verbal Memory task was completed by each participant. Participant then started walking on the treadmill at either a speed of 3.0 mph (4.8 km/h) for sedentary individuals or 3.5 mph (5.6 km/h) for active individuals with grade 0% (Hanson, 1984). This was followed by an increase in grade of 2% for every 2 mins with the speed remaining constant until targeted HR was reached. A heart rate (HR) monitor (POLAR®) was used to measure HR throughout the test and rating of perceived exertion (RPE) was done at the end of every 2 min stage. Exercise was stopped as soon as participant reaches targeted HR or requests to stop because of fatigue or any discomfort. Participant was then given time to cool down until HR reached or fell below 120 bpm and was allowed to take a break for approximately 1 min before proceeding with the second set of Verbal Memory Task. Upon completing the memory test, the participant was allowed to leave

SUMMARY:
Anxiety levels among the younger generation especially students have been increasing drastically in recent years. This severely affects a student's academics as previous studies have shown a strong correlation between high anxiety levels and poor working memory. Working memory, also known as short term memory is an important component in studying as it aids in holding important information needed to understand following information for a short period of time. This concerning phenomenon has drawn the attention of researchers to find solutions to this issue where recent studies have found physical exercise to contribute in the improvement of cognition which also includes working memory. Hence, the aim of this study is to compare the effects of low and high intensity exercises on working memory among students with high anxiety levels. Thirty female undergraduate students from UTAR with relatively high levels of anxiety will be conveniently sampled using Beck Anxiety Inventory. Participants will then be randomly allocated into 2 groups to undergo low and high intensity exercise on a treadmill according to Balke's Protocol. 2 memory assessments involving Verbal Memory Task will be conducted for each participant before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female students (Age group: 18-25 years)
* Participants with mild to severe anxiety levels (Score of >8)

Exclusion Criteria:

* Participants with Cardiorespiratory problems (e.g. Asthma, Congestive heart disorders) or severe Musculoskeletal problems that prevent them from carrying out any physical exercise or advised by personal physician not to.
* Participants that have had a recent head injury (recent 5 years)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Verbal Memory Task | baseline and 1 minutes
  Immediate effect of low and high intensity exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Tunku Abdul Rahman, Kajang, Selangor, Malaysia